CLINICAL TRIAL: NCT05933252
Title: A Pilot Clinical Trial to Determine the Feasibility of Administering an Electronic Tool to Assess Postoperative pAin, Nausea, and Vomiting in English or Spanish-Speaking Pediatric Patients With Neoplastic Conditions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Drug Abuse (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0097; NCI-2023-04990 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-06-19; First posted 2023-07-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Neoplastic Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented reality (AR) (Experimental): Augmented reality (AR)
  Participants will view the real world through a device's camera and application ("app") but adds virtual or digital characters and items to the image
  Interventions: Other: Augmented reality (AR)

INTERVENTIONS:
Other: Augmented reality (AR) — an app on an iPad every 15 minutes

SUMMARY:
The feasibility of using an electronic tool to measure pain, nausea, and vomiting after surgery in English or Spanish-speaking pediatric cancer patients.

DETAILED DESCRIPTION:
Primary Objective:

To determine the feasibility of administering an AR-based electronic tool to assess postoperative pain, nausea, and vomiting in English or Spanish-speaking pediatric patients with neoplastic conditions.

Secondary Objectives:

1. To evaluate the willingness to use the AR app,
2. To evaluate the time spent using the AR app (recorded in the study device),
3. To calculate the difference (delta) between pain and nausea intensity recorded from the app and those gathered by nursing personnel,
4. To evaluate app recorded responses to pain intensity,
5. To evaluate app recorded responses to nausea intensity,
6. To assess the frequency of vomiting,
7. To measure the length of stay in PACU (calculated from the EMR),
8. To determine the rate (number) of assessments completed,
9. To calculate PACU opioid use,
10. To calculate opioid use during hospitalization,
11. To assess the quality of life using the PedsQL Cancer Module survey responses (administered by the study team),
12. To evaluate patient/caregiver satisfaction following the PACU stay
13. To assess nursing experience with AR tool following patient discharge from PACU.

Exploratory Objectives:

1. To assess the primary/secondary outcomes for the English and Spanish-speaking patients separately.
2. To correlate pain-reported intensity to the analgesia nociception index (ANI).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 7-17 years old,
2. Able to provide assent, and a legal guardian able to provide informed consent
3. Current diagnosis of pediatric cancer or benign neoplasm,
4. Surgery with an estimated duration longer than 2 hours,
5. An expected prescription of opioids during the inpatient perioperative period
6. Demonstrate capacity to comprehend and interact with the game in English or Spanish.

Exclusion criteria:

1. Any concerns from the principal investigator or primary team about the use of the app,
2. Inability or refusal from the parents to provide written informed consent.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Activation and use of the technology (YES versus NO) | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Juan Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT05933252/ICF_000.pdf